CLINICAL TRIAL: NCT04243200
Title: Effect of Implementing an Ambulance Clinician Delivered Hypoglycaemia Intervention ('Hypos Can Strike Twice') on Repeat Ambulance Calls, Attendances and Transportation to Hospital: Non-randomised Stepped Wedge and Process Evaluation
Brief Title: Ambulance 'Hypos Can Strike Twice' Study
Acronym: Ambu-HS2
Status: Completed | Type: Observational
Sponsor: University of Lincoln (Other)
Responsible Party: Sponsor
Other Study IDs: 191202
Record Dates: First submitted 2020-01-23; First posted 2020-01-28 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-04

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Analyses of repeat ambulance calls and costs: For our analyses of repeat ambulance calls and costs we will use routine anonymised data from routine call-and-dispatch and clinical records data from EMAS for 12 months before the intervention was first introduced (September 2017) to at least 6 months after the final step of the introduction in April 2019, i.e. October 2019. This is likely to involve the analysis of an estimated 11916 cases so that we can implement a stepped wedge (non-randomised control)design .
  Interventions: Other: Hypos can strike twice
- Survey of patients receiving intervention: We will survey about 447 patients who received the intervention in order to obtain data from a sample of n=96
  Interventions: Other: Hypos can strike twice
- Survey of ambulance staff: We will send out surveys/questionnaires to all front-line ambulance staff (n=approximately 600)
- Qualitative interviews of staff: We will sample 10-15 staff for qualitative interviews.
- Qualitative interviews of patients: We will sample 10-15 patients for qualitative interviews
  Interventions: Other: Hypos can strike twice

INTERVENTIONS:
Other: Hypos can strike twice — The "Hypos can strike twice" intervention involves ambulance staff providing treatment to patients experiencing hypos and advising them to access follow-up care by their GP/specialist diabetes team. This is backed up by giving patients a "Hypos can strike twice" information booklet which they can read when they recover.
  Groups: Analyses of repeat ambulance calls and costs; Qualitative interviews of patients; Survey of patients receiving intervention

SUMMARY:
This study will assess the effectiveness the "Hypos can strike twice" intervention on people with diabetes experiencing hypoglycaemia (or "hypo", meaning low blood sugar). The intervention should help prevent recurrence of "hypos", improve patients' future health, reduce calls to ambulance services and thus reduce NHS pressures and costs.

Hypoglycaemia affects increasing numbers of people with diabetes. It is a side effect of treatment with insulin or certain tablets, where blood glucose (sugar) falls causing the brain to malfunction. In mild cases this can lead to sweating, drowsiness and confusion; in more severe cases, coma can occur needing medical assistance for recovery, and if prolonged can be fatal. It results in 1% of calls to ambulance services.

The "Hypos can strike twice" intervention involves ambulance staff providing treatment to patients experiencing hypos and advising them to access follow-up care by their GP/specialist diabetes team. This is backed up by giving patients a "Hypos can strike twice" information booklet which they can read when they recover.

Universities of Lincoln and Leicester are working with East Midlands Ambulance Service NHS Trust and patient groups on this study. The "Hypos can strike twice" intervention has now been implemented by ambulance services in Leicester, Northamptonshire, Nottinghamshire, Derbyshire and Lincolnshire from October 2018-May 2019.

The investigators will analyse data from the ambulance services before, during and after the introduction of the 'Hypos can strike twice' intervention to evaluate the effect of the intervention on repeat ambulance calls and attendances for hypoglycaemia and the costs and consequences of implementing it. The investigators will also interview/survey ambulance staff who provided the intervention and patients who received it, to understand how and why it works (or does not) and how, if it works, it could be scaled up over a larger geographical area. The duration of this study is 1 year.

DETAILED DESCRIPTION:
Research question

What is the effect on repeat ambulance calls and attendances for hypoglycaemia and what are the costs and consequences of implementing the 'Hypo's can strike twice' intervention to patients with diabetes and hypoglycaemia attended by East Midlands Ambulance Service NHS Trust in the East Midlands region of the UK?

Background

Severe hypoglycaemia (defined as cognitive impairment severe enough to require external assistance for recovery) frequently requires an ambulance resulting in Emergency Department attendance or hospital admission. Severe hypoglycaemia constitutes around 1% of 1.7 million emergency ambulance calls in England and Scotland resulting in 100 thousand paramedic attendances and estimated costs in England of £13.6 million annually. Hypoglycaemia is associated with adverse consequences including higher mortality, morbidity and health service costs due to hospital attendance/admission. It is also frightening for both patients and relatives and impairs quality of life and productivity, leading to poor long term control.

Aims and objectives

Aim: To evaluate the effect of implementing the 'Hypo's can strike twice' intervention to patients with diabetes and hypoglycaemia attended by East Midlands Ambulance Service NHS Trust in the East Midlands region. "Hypos can strike twice" is a complex intervention involving ambulance staff providing treatment and advice to people who have had a hypoglycaemic attack to access follow-up care by the GP or specialist diabetes team as detailed in national ambulance (JRCALC) clinical guidelines supported by the provision of a "Hypos can strike twice" booklet which the patient can read when they are fully recovered from the cognitive and other effects of the hypoglycaemic episode.

Objectives

To investigate the effect of implementing the 'Hypo's can strike twice' on:

1. Repeat ambulance calls and attendances for hypoglycaemia
2. Recorded referrals to an appropriate healthcare professional (e.g. GP, nurse).
3. Completed care bundle for hypoglycaemia (proportion of patients with all of blood glucose recorded before treatment, blood glucose recorded after treatment and treatment given for hypoglycaemia.
4. Costs of implementation 'Hypo's can strike twice' intervention vs costs of health service resource use.
5. To conduct a process evaluation to explore how 'Hypo's can strike twice' exerts its effects and can be scaled up if effective by understanding implementation, mechanisms of impact, and contextual factors using interviews and surveys

Methods

Non-randomised stepped wedge design with mixed-methods process evaluation.

ELIGIBILITY:
Inclusion criteria:

Patients: Adults aged 18 years+ with diabetes experiencing hypoglycaemia needing an ambulance service response. Hypoglycaemia for this study was identified as a 'clinical impression' of 'hypoglycaemia' or 'diabetic problem'. Hypoglycaemia may also be identified according to ambulance guidelines1 as any blood glucose less than 4mmol/L.

Clinicians: Ambulance staff providing treatment and advice to people who have had a hypoglycaemic attack.

Exclusion Criteria:

Patients: Children under the age of 18 years.

Clinicians: Ambulance staff providing treatment and advice for incidents other than hypoglycaemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients needing an ambulance for hypoglycaemic events and ambulance staff attending these events.
Sampling Method: Non-Probability Sample
Enrollment: 5015 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Repeat ambulance calls and attendances for hypoglycaemia within 14 days. | 14 days from initial ambulance attendance
  as stated above

SECONDARY OUTCOMES:
To assess whether the "Hypos can strike twice" intervention can reduce repeat ambulance calls and attendance for hypoglycaemia within 30 and 90 days. | within 30 and 90 days from initial ambulance attendance
  as stated above

CONTACTS AND LOCATIONS:
Overall Officials: Niro Siriwardena, Principal Investigator — University of Lincoln, UK
Locations (1):
- Community and Health Research Unit, University of Lincoln, Lincoln, Lincolnshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Laparidou D, Botan V, Law GR, Rowan E, Smith MD, Brewster A, Spaight R, Mountain P, Dunmore S, James J, Roberts L, Khunti K, Siriwardena AN. People with diabetes and ambulance staff perceptions of a booklet-based intervention for diabetic hypoglycaemia, "Hypos can strike twice": a mixed methods process evaluation. BMC Emerg Med. 2022 Feb 8;22(1):21. doi: 10.1186/s12873-022-00583-y. PMID 35135499